CLINICAL TRIAL: NCT04513639
Title: The Relapse from MRD Negativity As Indication for Treatment (REMNANT) Study
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); Haukeland University Hospital (Other); University Hospital of North Norway (Other); University Hospital, Akershus (Other); Helse Stavanger HF (Other Government); Førde Central Hospital (Other); Sorlandet Hospital HF (Other Government); Nordlandssykehuset HF (Other); The Hospital of Vestfold (Other); Helse Nord-Trøndelag HF (Other); Alesund Hospital (Other); Sykehuset Ostfold (Other)
Responsible Party: Principal Investigator, Fredrik Hellem Schjesvold, Head of Oslo Myeloma Center, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMC01/19
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental): Patients will be followed with MRD assessment every 4 month and start 2.L treatment at loss of MRD negative complete response.
  Interventions: Drug: Early treatment of relapse with carfilzomib, dexamethasone, daratumumab
- Arm B (Active Comparator): Patients will be followed up by standard criteria and start 2.L treatment at progressive disease.
  Interventions: Drug: Standard treatment of relapse with carfilzomib, dexamethasone, daratumumab

INTERVENTIONS:
Drug: Early treatment of relapse with carfilzomib, dexamethasone, daratumumab — Second line treatment will start at MRD reapperance
  Other Names: DKd
  Arms: Arm A
Drug: Standard treatment of relapse with carfilzomib, dexamethasone, daratumumab — Second line treatment will start at progressive disease
  Other Names: DKd
  Arms: Arm B

SUMMARY:
The REMNANT study will evaluate whether treating minimal residual disease (MRD) relapse after first line treatment prolongs progression free survival and overall survival for myeloma patients versus treating relapse after first line treatment at progressive disease. To establish a homogenous group of MRD negative patients after first line treatment including autologous stem cell transplantation, patients are enrolled at diagnosis and treated with Norwegian standard of care first line treatment. MRD negative patients will move on to the randomized part.

DETAILED DESCRIPTION:
391 patients with newly diagnosed multiple myeloma eligible for high dose therapy with autologous stem cell support will be included in the phase II part of the study and receive standard of care first line treatment according to Norwegian national guidelines; bortezomib- lenalidomide - dexamethasone for 4 pre-transplant induction and 4 post-transplant consolidation cycles (all 21-d cycles). After induction patients will undergo tandem or single ASCT, depending on toxicity and response to first ASCT. The primary endpoint of the phase 2 part of the study is the number of patients who achieve MRD negative (Euroflow NGF 10 -5 ) complete response 30-45 days post consolidation. Patients (176) achieving MRD negative complete response will be randomly assigned in a 1:1 ratio to receive second line treatment at MRD reappearance (arm A) or at progressive disease as defined by the IMWG criteria (arm B). Randomization will be stratified by R-ISS stage at diagnosis and single vs tandem ASCT. Patients in arm A will be followed with MRD assessment every 4 month and start second line treatment at loss of MRD negative CR. Patients in arm B will be followed up by standard criteria and start second line treatment at progressive disease. Both arms will receive the same 2.L treatment; carfilzomib - dexamethasone - daratumumab. (all 28-d cycles) Second line treatment will continue until disease progression, unacceptable AEs or patient withdrawal. In arm A MRD Euroflow will be assessed after 6 and 18 months of 2L therapy. In arm B MRD Euroflow will be assessed if >CR is achieved but not before 6 months of 2 L therapy, and again after 12 consecutive months.

ELIGIBILITY:
Inclusion Criteria part one:

* Each patient must meet all of the following inclusion criteria to be enrolled in the study:

  1. Patient with newly diagnosed multiple myeloma (IMWG criteria) eligible for high-dose therapy and ASCT.
  2. Patient must be >18 and < 75 years of age at the time of signing the informed consent
  3. Must have measurable disease as defined by the International Myeloma Working Group; serum monoclonal paraprotein (M-protein) level > 10 g/L or light chain multiple myeloma without measurable disease in the serum; serum immunoglobulin FLC > 100 mg/L and abnormal serum immunoglobulin kappa lambda FLC ratio.
  4. Voluntary written informed consent
  5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2. ECOG 3 can be enrolled if caused by myeloma.
  6. Patient must be willing and able to adhere to the study protocol visit schedule and other protocol requirements.
  7. Female of childbearing potential (FCBP) must have a confirmed negative serum pregnancy test within 7 days prior to inclusion.
  8. FCBP and male subject who are sexually active with FCBP must agree to use highly effective concomitant methods of contraceptive during the study and for at least 28 days following the last study drug dose. Male subjects must use contraception and refrain from donating sperm for at least 28 days after the last dose of lenalidomide according to Pregnancy Prevention Plan (Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information).

     Inclusion Criteria part two:
* Each patient must meet all of the following inclusion criteria to be enrolled in the study

  1. Patient must be MRD negative measured by Euroflow NGF after 1.L therapy. The cutoff for inclusion into part 2 will be 100 PC per 10 mill. nucleated cells monitored in BM.
  2. Has received 1.L treatment in part 1 of the study.
  3. ECOG performance status score 0, 1 or 2

Exclusion Criteria part one:

1. Received more than one cycle of induction treatment for multiple myeloma.
2. Patient with ongoing or active systemic infection, active hepatitis B or C virus infection or known human immunodeficiency virus (HIV) positive
3. Concurrent medical or psychiatric condition or disease that is incompatible to HDM and ASCT or that will likely result in reduced study compliance and reduce ability to follow study procedures, or that in the opinion of the investigator, would constitute a hazard for participating in this study.
4. No active malignancy with a lower life expectancy than myeloma
5. Female patient who have a positive serum pregnancy test during the screening period.
6. Female patient who is lactating during the screening period but are not willing to stop lactating prior to the first treatment cycle starts.
7. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.

Exclusion Criteria part two:

1. No active malignancy with a lower life expectancy than myeloma
2. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2020-08-27 (Actual); Primary Completion 2031-06-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 10 years
  Median PFS of Arm A (MRD guided) vs Arm B (PD guided) defined as the time from randomization to disease progression or death due to any cause following 2.L treatment.
Overall survival (OS) | 11 years
  Median OS of Arm A vs Arm B (MRD guided) defined as the time from randomization to death of any cause following 2.L treatment.
Minimal residual disease negativity after first line treatment | 30-45 days post consolidation
  The number of participants who achieve MRD negativity measured by Euroflow NGF at 30-45 after consolidation therapy has ended

SECONDARY OUTCOMES:
Time-to-next treatment | 10 years
  Time from end of first line treatment to start of 3.L therapy
Minimal residual disease negativity during second line treatment | 6 months after starting second line treatment
  The proportion of patients who achieve MRD negativity during 2.L treatment, monitored by MRD Euroflow NGF at 6 and 18 months in arm A and after achieving CR in arm B (first MRD testing after 6 months).
Health-related quality of life (HRQOL) | 10 years
  Patient reported outcome HRQOL forms will be filled out by patients at defined time points during the study and finally at relapse after 2.L therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Schjesvold, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (13):
- Norway (13):
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Nordland Hospital Bodø, Bodø
  - Sykehuset Ostfold, Fredrikstad
  - Førde Central Hospital, Førde
  - Sørlandet Hospital Kristiansand, Kristiansand
  - Levanger Hospital, Levanger
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - Helse Stavanger HF, Stavanger
  - University Hospital North Norway, Tromsø
  - St. Olavs Hospital, Trondheim
  - The Hospital of Vestfold, Tønsberg

IPD SHARING:
Plan to Share IPD: No